CLINICAL TRIAL: NCT04902794
Title: Light Emitting Diode in the Treatment of Genitourinary Syndrome of Menopause: Randomized Controlled Clinical Trial
Brief Title: Light Emitting Diode in the Treatment of Genitourinary Syndrome of Menopause
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Patricia Lordelo (Other)
Collaborators: University of Messina (Other)
Responsible Party: Sponsor-Investigator, Patricia Lordelo, Principal Investigator, Centro de Atenção ao Assoalho Pélvico
Organization: Centro de Atenção ao Assoalho Pélvico (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1201-2342
Record Dates: First submitted 2021-05-20; First posted 2021-05-26 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Atrophy;Vaginal
Keywords: Phototherapy; Menopause; Women

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light Emitting Diode (Experimental): Light Emitting Diode in the Treatment of Menopause Genitourinary Syndrome
  Interventions: Device: Light Emitting Diode
- Light Emitting Diode Sham (Sham Comparator): Light Emitting Diode device Sham - turned off
  Interventions: Device: Sham Light Emitting Diode

INTERVENTIONS:
Device: Light Emitting Diode — Blue light-emitting diode applied to the female genital region for eight minutes, for five sessions, one per week
  Arms: Light Emitting Diode
Device: Sham Light Emitting Diode — Sham Blue light-emitting diode turned off applied to the female genital region for eight minutes, for five sessions, one per week
  Arms: Light Emitting Diode Sham

SUMMARY:
Introduction: The genitourinary menopause syndrome (MMS) affects 50% of postmenopausal women and, due to a decrease in hormone levels, triggers functional changes in the vagina and vagina, and impairment of quality of life and sexual function. Objective: To test the hypothesis that the 405 nm light emitting diode in the treatment of vulvovaginal atrophy is safe and effective, by reducing the symptomatology of the disease and histological alteration of the tissue. Methods: This is a pilot study in 10 volunteers with SGM, followed by a randomized, blinded trial in a sample of 58 individuals that will be performed at the Pelvic Floor Care Center (CAAP). Menopausal women up to 65 years of age and with clinical signs and symptoms of vulvovaginal atrophy syndrome (vaginal dryness and irritation, pruritus, pain or discomfort in intercourse, bleeding after sexual intercourse) and who voluntarily participate in the study will be included. Will be excluded from the study the patients in hormonal replacement for less than 6 months, diagnosis of vaginal infection, use of pacemaker, pregnant women, those who have performed Oophorectomy or presented ovarian cancer, difficulty understanding the proposed instruments and patients with chronic neurological degenerative diseases. Three 405 nm light emitting diode (LED) sessions will be performed, with a seven days interval between them. In the clinical trial, the study group will perform kinesiotherapy and LED.

The control group will perform kinesiotherapy and the LED will be turned off. Data collection will be performed initially and after the sessions through self-administered questionnaires containing socio-demographic and clinical information, Medical Outcomes Study 36, Short-Form Health Survey (SF-36), Female Sexual Function Index (FSFI) - Female Version (QS-F), Female Genital Self-Image Scale - 7 (FGSIS-7). At the end of treatment, the visual analog scale and Likert scale will be used to measure the individual's satisfaction. Expected results: The 405nm LED in the vaginal canal is expected to be safe and effective for SGM.

ELIGIBILITY:
Inclusion Criteria:

* menopausal women up to 65 years of age
* presence of clinical signs and symptoms of Menopause Genitourinary Syndrome :dryness and irritation of the vagina, pruritus, pain or discomfort in sexual intercourse, bleeding after sexual intercourse
* voluntarily participate in the research.

Exclusion Criteria:

* patients undergoing hormone replacement for less than 6 months
* diagnosis of vaginal infection
* difficulty in understanding the proposed instruments
* patients with chronic neurological degenerative diseases.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Vaginal maturation index | Change from baseline at 3 months
  Cytological vaginal will be collected at one third lower lateral vaginal wall and quantified superficial, intermediate and basal cells to calculate vaginal maturation index
Female Sexual Function Index (FSFI) - Female Version (QS-F) | Change from baseline at 3 months
  Measure of quality of sex life. Full Scale Score Range 2-36 - The higher final score, better is the sexual function

SECONDARY OUTCOMES:
Vaginal pH | Change from baseline at 3 months
  pH indicator tape
Urinary symptoms | Change from baseline at 3 months
  International Consultation on Incontinence Questionnaire - Short Form (ICIQ Questionary Short Form)-Scoring scale: 0-21 (lower values means better quality of life)
Visual analog scale | Change from baseline at 3 months
  Stratification between 0 and 10 (few symptoms to severe symptoms)
Female Genital Self-Image Scale - 7 (FGSIS-7) | Change from baseline at 3 months]
  Measure of quality of sex life. Scores between 7-28 (higher scores indicate better self-image)
Likert scale | Change from finished treatment and 3 months after
  Satisfaction with the treatment measured between 1 and 5 ( not at all happy with the treatment -very happy with the treatment)
Sexual Quotients Female Version (QS-F) | Change from baseline at 3 months
  Female sex life domain. Scores between 0-100 (higher scores indicate better sex life) Scores between 82-100 score: excellent, 62-80 score: regular, 42-60 score: unfavorable, 22-40 score: regular, 0-20 score: bad
SF-36 | Change from baseline at 3 months
  Short Form health survey 36 questionnaire, (0-100) - lower values means worse quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Patrícia Lordelo, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No